CLINICAL TRIAL: NCT05906342
Title: Investigating the Effect of Acute Fat Ingestion on Glucose Metabolism in Young Healthy Adults: a Dose Response Study
Brief Title: Dose Response Relationship Between Fat Ingestion and Metabolism
Acronym: AFDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Kirsten Bell, Principal Investigator, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16153
Record Dates: First submitted 2023-03-11; First posted 2023-06-15 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Glucose Tolerance Impaired
Keywords: High-fat; Glucose; Insulin; Metabolism; Nutrition
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Each participant will be required to consume four breakfast meals (containing 20, 40, 60, or 80% energy from fat) in a randomized order with a washout period between meals
Who Masked: Participant, Investigator
Masking Description: Participants and investigators will not know the fat quantity of the meal that is being consumed or the order in which the meals are provided to the participant. A non-investigator member of the research team will be responsible for creating the meals and keeping track of which meals are being consumed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 20% fat meal (Experimental): This meal will contain 15 kcal/kg of body weight and consist of 20% fat, 65% carbohydrates, and 15% protein.
  Interventions: Other: 20% fat meal
- 40% fat meal (Experimental): This meal will contain 15 kcal/kg of body weight and consist of 40% fat, 45% carbohydrates, and 15% protein.
  Interventions: Other: 40% fat meal
- 60% fat meal (Experimental): This meal will contain 15 kcal/kg of body weight and consist of 60% fat, 25% carbohydrates, and 15% protein.
  Interventions: Other: 60% fat meal
- 80% fat meal (Experimental): This meal will contain 15 kcal/kg of body weight and consist of 80% fat, 5% carbohydrates, and 15% protein.
  Interventions: Other: 80% fat meal

INTERVENTIONS:
Other: 20% fat meal — Provided to participants once throughout duration of study, contains 20% fat
  Arms: 20% fat meal
Other: 40% fat meal — Provided to participants once throughout duration of study, contains 40% fat
  Arms: 40% fat meal
Other: 60% fat meal — Provided to participants once throughout duration of study, contains 60% fat
  Arms: 60% fat meal
Other: 80% fat meal — Provided to participants once throughout duration of study, contains 80% fat
  Arms: 80% fat meal

SUMMARY:
The goal of this clinical trial is to compare features of metabolism in healthy, young adults after they consume four meals of differing fat quantity. The main question this trial aims to answer is how does increasing fat quantity impact glucose tolerance, glucose and insulin metabolism, and hormones involved in hunger. Participant will consume four meals consisting of either 20, 40, 60, or 80% energy from fat.

DETAILED DESCRIPTION:
The long-term consumption of high-fat foods can lead to unhealthy changes in the functioning of the body, giving rise to metabolic diseases such as type 2 diabetes. Similarly, short-term high-fat diets have also been shown to disrupt how the body performs but there is a lack of information regarding how a single high-fat meal can disrupt metabolism. Comparing meals of different fat quantity, without changing the overall energy intake (calories), will help us understand the short-term effect of fat ingestion on the functioning of the body and whether increasing the amount of fat in a meal is related to the level of dysfunction in the body. Therefore, the investigators will provide participants with four meals of varying fat quantity and in the period following the meal, the investigators will take blood samples to determine any changes that occur in the body in response to different levels of fat.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 and 30.0 kg/m2
* Weight stable for the past 6 months (± 2kg)
* VO2max values within a below average to above average range (38-50 mL/kg and 35-47 mL/kg for 18-25 year old males and females respectively. 35-48 mL/kg and 34-45 mL/kg for 26-35 year old males and females respectively)
* Fasting blood glucose <6.0 mM
* Resting blood pressure <140/90 mmHg
* Taking second generation oral contraceptives (females only)

Exclusion Criteria:

* Smoking
* Diabetes, cancer, or other metabolic disorders
* Cardiac or gastrointestinal problems
* Infectious disease
* Barium swallow or nuclear medicine scan in the previous 3 weeks
* Follow a strict vegan diet
* Pregnant or breastfeeding (females only)
* Diagnosis of polycystic ovary syndrome (females only)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Glucose tolerance | Two hours (taking place following the 4-hour postprandial period)
  A 2-hour intravenous glucose tolerance test will be performed 4-hours after meal consumption

SECONDARY OUTCOMES:
Glucose and lipid metabolites | During the 4-hour postprandial period
  Postprandial availability of glucose (mM)
Glucose and lipid metabolites | During the 4-hour postprandial period
  Postprandial availability of insulin (µIU/mL)
Glucose and lipid metabolites | During the 4-hour postprandial period
  Postprandial availability of total cholesterol (mmol/L)
Glucose and lipid metabolites | During the 4-hour postprandial period
  Postprandial availability of low-density lipoprotein (mmol/L)
Glucose and lipid metabolites | During the 4-hour postprandial period
  Postprandial availability of high-density lipoprotein (mmol/L)
Glucose and lipid metabolites | During the 4-hour postprandial period
  Postprandial availability of non-esterified fatty acids (mmol/L)

OTHER OUTCOMES:
Hunger hormones | During the 4-hour postprandial period
  Postprandial concentration of ghrelin (pmol/L)
Hunger hormones | During the 4-hour postprandial period
  Postprandial concentration of leptin (pmol/L)
Hunger hormones | During the 4-hour postprandial period
  Postprandial concentration of adiponectin (pmol/L)

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Ivor Wynne Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to other researchers